CLINICAL TRIAL: NCT06450171
Title: Evaluation of Multi-Cancer Early Detection Testing in a High-Risk Population: The INFORM Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Elizabeth ODonnell, Sponsor Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 24-070
Record Dates: First submitted 2024-06-04; First posted 2024-06-10 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Cancer Predisposition Syndrome; Predisposition, Genetic
Keywords: Cancer Predisposition Syndrome; Predisposition, Genetic
MeSH Terms: conditions — Genetic Predisposition to Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Galleri MCED Test (Experimental): Participants will be enrolled and will complete:
  * Baseline questionnaires and blood test.
  * Post-test questionnaires.
  * Follow-up assessments for a negative GRAIL Galleri test include recommended cancer screenings and a follow up phone call with study staff 1 year after the GRAIL Galleri blood test.
  * Follow-up assessments for a positive GRAIL test may include clinic visits, lab tests with additional blood work-ups, biopsies, surgical procedures, or imaging assessments such as ultrasound, Computed Tomography (CT) scans, or an Magnetic Resonance Imaging (MRI) scans.
  * If cancer status is confirmed, participants will complete a post-diagnostic questionnaire.
  Interventions: Other: GRAIL Galleri Test

INTERVENTIONS:
Other: GRAIL Galleri Test — A multi-cancer early detection (MCED) blood test.

SUMMARY:
The purpose of this research study is to evaluate the possible benefits and harms of screening with an investigational blood test designed to detect many types of cancer early.

The name of the screening blood test being studied is:

-GRAIL Galleri test

DETAILED DESCRIPTION:
This is a prospective, interventional study to assess the use of the GRAIL's Galleri multi-cancer early detection (MCED) Test, an investigational blood test designed to detect many types of cancer, for participants that are considered at slightly higher than average risk of developing certain types of cancers. The test looks for small pieces of genetic material called deoxyribonucleic acid (DNA) in the blood that may indicate the presence of cancer.

The research study procedures include screening for eligibility, blood tests, questionnaires, and clinic visits.

Participation in this research study is expected to last up to 3 years.

It is expected that about 1,000 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria Group 1- Cancer Predisposition Syndrome:

* Age ≥ 22 for patients with TP53 germline pathogenic variants, age ≥ 35 for all other variants in cancer predisposing genes
* Germline genetic testing revealed pathogenic germline variants in cancer predisposing genes (list of genes typically tested listed in pre-screening document)
* Individuals with a clinically based diagnosis of a Cancer Predisposition Syndrome (examples, neurofibromatosis, Fanconi Anemia, Ataxia-Telangiectasia)

Inclusion Criteria Group 2 - Familial Risk:

* Age ≥ 45
* Adults with family history suggestive of elevated cancer risk as defined by any the criteria below, who do not fall into Group 1:

  * ≥ 1 first or second degree relative on same side of the family with:

    * Breast, colon, gastric, endometrial, kidney cancer at or before age 50
    * Triple negative breast cancer (any age)
    * Male breast cancer (any age)
    * Ovarian, pancreatic, sarcoma cancer (any age)
    * Neuroendocrine cancer or tumors (any age)
    * Metastatic prostate cancer (any age)
    * Multiple primary cancers (example bilateral breast cancer)
  * ≥ 2 first or second degree relative on same side of the family (any combination is acceptable) with breast or prostate cancer at any age

Exclusion Criteria:

* Individuals diagnosed with invasive malignancy within 3 years of enrollment
* Have had a blood-based multi-cancer screening test within last year
* Individuals with evidence of symptomatic or active cancer requiring active therapeutic intervention at the time of participation (hormone therapy for breast/prostate cancer is considered acceptable and will not preclude participation)
* Individuals in Group 2 whose family history of cancer was the result of a germline mutation in a cancer predisposing gene and who have tested negative for that same familial germline mutation
* Individuals in Group 2 whose family history of cancer is sex-specific and who is a different sex than the proband with cancer (e.g., a male with a family history of endometrial or ovarian cancer would not be eligible)
* Individuals in process of being evaluated for clinical suspicion of cancer
* Individuals who have undergone a cancer risk-reducing surgery for hereditary cancer risk (e.g., mastectomy)

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-09-27 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Cancer Detection Rate | Up to 2 years
  Descriptive statistics will be used to summarize the number and types of cancers diagnosed by GRAIL Galleri MCED testing.

SECONDARY OUTCOMES:
Stage of Invasive Cancer Diagnosis | Up to 2 years
  Descriptive statistics will be used to summarize the stages of invasive cancer that are diagnosed by GRAIL Galleri MCED testing and assessed by medical record review.
Positive Predictive Value At 12 Months | At 12 months
  Positive Predictive Value is defined as the proportion of participants with cancer diagnosis out of all participants with "signal detected" on GRAIL Galleri MCED test results.
Positive Predictive Value at 24 Months | At 24 months
  Positive Predictive Value is defined as the proportion of participants with cancer diagnosis out of all participants with "signal detected" on GRAIL Galleri MCED test results.
Time to Diagnostic Resolution | Calculated from the date of return of screening results (up to 4 weeks from baseline) until up to 24 months post screening
  Defined as the time required to achieve diagnostic resolution following a "signal detected" GRAIL Galleri MCED test result.
Test Type Utilization to Diagnostic Resolution | Up to 24 months
  Per participant the count of the number and types of diagnostic tests required to achieve diagnostic resolution following a "signal detected" GRAIL Galleri MCED test result.
Change in Participant Anxiety | Up to 24 months
  Changes in anxiety following the GRAIL Galleri MCED test result and assessed by the Patient-Reported Outcome Measurement Information System (PROMIS) Emotional Distress Anxiety - Short Form 6a, which is a 6 item survey that is rated on a 5-point Likert scale with answers ranging from "Never" to "Always". The range of scoring is from 6 to 30 with higher scores indicating greater severity of anxiety.
Change in Participant Health-related Quality of Life | Up to 24 months
  Changes in health-related quality of life following the GRAIL Galleri MCED test result and assessed by PROMIS Scale v1.2 - Global Health, a 10 item survey that is rated on a 5-point Likert scale with answers ranging from "Excellent/Completely/Never/None" to "Poor/Not at all/Always/Very Severe" and includes a pain average question rated on a scale of 0 "No Pain" to 10 "Worst Pain Imaginable." The range of scoring is from 9 to 45 with higher scores indicating higher quality of life.
Cost of Follow-up Testing | Up to 24 months
  Defined as the dollar cost, per participant, of follow-up testing to achieve diagnostic resolution following a "signal detected" GRAIL Galleri MCED test result.
Institutional Reimbursement of Follow-up Testing | Up to 24 months
  Defined as the dollar cost, per participant, of the institutional reimbursement of follow-up testing to achieve diagnostic resolution following a "signal detected" GRAIL Galleri MCED test result.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth ODonnell, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu